CLINICAL TRIAL: NCT06979310
Title: The Comparative Effectiveness Evaluation of the Impact of Digital Education Via Text Message Versus Multimedia Modules on Caregiver Knowledge
Brief Title: The Comparative Effectiveness Evaluation of the Impact of Digital Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00115965; 1R21CA284299-01 (NIH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- text-based education messages only (Active Comparator)
  Interventions: Other: text-based education messages only
- in-clinic tablet-based multimedia education only (Active Comparator)
  Interventions: Other: in-clinic tablet-based multimedia education
- both text-based and tablet-based digital education strategies (Active Comparator)
  Interventions: Other: text-based education messages only; Other: in-clinic tablet-based multimedia education
- standard of care provider led education (Active Comparator)
  Interventions: Other: standard of care provider led education

INTERVENTIONS:
Other: text-based education messages only — Participants will receive text-based education messages
  Arms: both text-based and tablet-based digital education strategies; text-based education messages only
Other: in-clinic tablet-based multimedia education — Participants will receive tablet-based multimedia education in clinic
  Arms: both text-based and tablet-based digital education strategies; in-clinic tablet-based multimedia education only
Other: standard of care provider led education — Participants will receive standard of care education from their provider
  Arms: standard of care provider led education

SUMMARY:
This study is being conducted to determine how best to educate caregivers about cancer and its treatment. When caregivers are well-informed, they are more confident in supporting their child through treatment, which can improve treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* a known pediatric cancer diagnosis
* Adult caregivers of children with cancer (<18yo) at time of new patient registration
* Ability to understand and speak Swahili
* If illiterate, availability of a household member who can read Swahili
* Be able to access the messages

Exclusion Criteria:

* any potential participant who is unable to access messages will also be excluded.
* Non cancer pediatric diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment abandonment rate. | 6 months
  All analyses estimating efficacy of the intervention will be based on intention-to-treat principles, whereby participants will be analyzed according to their randomization assignment, irrespective of whether they complied with the intervention.

SECONDARY OUTCOMES:
Caregiver knowledge | Baseline, 6 months
  Caregiver knowledge will be assessed by a 10-question multiple choice survey testing core knowledge on childhood cancer
Caregiver attitudes | Baseline, 6 months
  Caregiver attitudes will be assessed by a version of the Swahili Cataldo Cancer Stigma Scale (CASS) previously modified to target childhood cancer stigma and validated for use in Tanzania by the current study team. Responses are rated using a four-point Likert scale to evaluate the caregivers attitude towards the statements (ranging from 1=strongly disagree; 4=strongly agree)
Perceived behavior control | Baseline, 6 months
  Perceived behavioral control will be assessed using a modified Swahili Generalized Self -Efficacy survey, adapted for use to evaluate caretaker perceived ability to complete therapy as the behavior measured. This is a 12 question item survey with a 5 point Likert scale (1=Not at all confident to 5=Extremely confident).
Caregiver intention | Baseline, 6 months
  Behavior intention will be assessed using a 3-question validated measure of intention translated into Swahili to determine caregiver's intention to complete therapy, with scaled response options from 1 to 7, from "strongly disagree/ very unlikely" to "strongly agree/ very likely."

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Schroeder Principal Investigator, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No
All enrolled participants will be assigned a study identification number (ID) to help protect their identity during data collection and analysis. Only study IDs will be used to identify participants' medical record data, survey and interview responses.